CLINICAL TRIAL: NCT02043990
Title: Patient Ventilator Interaction During Non-invasive Ventilation Delivered With Neurally Adjusted Ventilatory Assist (NAVA-NIV) in Infants
Brief Title: Adjusted Ventilatory Assist (NAVA-NIV) in Infants: Short-term Physiological Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCHIDINI2013
Record Dates: First submitted 2013-04-28; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Acute Respiratory Failure
Keywords: NAVA; noninvasive ventilation; infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Noninvasive NAVA Ventilation (Experimental): Noninvasive NAVA Ventilation versus conventional noninvasive Pressure Support Ventilation
  Interventions: Device: Noninvasive NAVA ventilation

INTERVENTIONS:
Device: Noninvasive NAVA ventilation — Noninvasive NAVA Ventilation versus conventional noninvasive Pressure Support Ventilation

SUMMARY:
Neurally Adjusted Ventilatory Assist (NAVA) is a new form of partial support wherein the machine applies positive pressure throughout inspiration in proportion to the electrical activity of the diaphragm (EAdi), as assessed by trans-esophageal electromyography. To test the hypothesis that NAVA could provide better patient-ventilator synchrony during NIV delivered by nasal-facial mask as compared to conventional flow-triggered PSV in infants with Acute Respiratory Failure.

DETAILED DESCRIPTION:
Neurally Adjusted Ventilatory Assist (NAVA) is a new form of partial support wherein the machine applies positive pressure throughout inspiration in proportion to the Electrical Activity of the diaphragm (EAdi), as assessed by trans-esophageal electromyography. Because ventilator functioning and cycling are under control of the patient's respiratory drive and rhythm, NAVA has the potential to enhance patient-ventilator interaction ensuring synchrony and minimizing the risk of over-assistance. A high incidence of asynchrony events has been demonstrated to have a significant clinical impact by favouring weaning failure and longer duration of mechanical ventilation.

NAVA has been implemented safely in animals, in healthy volunteers and in critically ill adults and has been shown to improve patient-ventilator synchrony, to limit excessive airway pressure and tidal volume, and to unload the respiratory muscles in tracheally intubated patients.

Moreover NAVA was found to be effective in delivering non-invasive ventilation (NIV) even when the interface was excessively leaky (75% leak) with reduced positive end-expiratory pressure. With these conditions, NAVA was able to unload the respiratory muscles and preserve gas exchange, while maintaining synchrony to respiratory demand. To date, no data exist on the use of NAVA in infants during noninvasive ventilation. The aim of this physiological study is to compare patient-ventilator interaction in infants receiving NIV by NAVA and Pressure Support Ventilation (PSV).

ELIGIBILITY:
Inclusion Criteria:

* Infants aging > 1 month and < 2 yrs
* ARF (PaO2/FiO2 < 300 mmHg)
* Accessory muscle recruitment
* Respiratory Rate more than 2 SD related to age
* Intact neuromuscular pathway to the diaphragm

Exclusion Criteria:

* Hemodynamic instability
* Facial Surgery
* Reduction in airway protection
* Coma
* Contraindication to insert the nasogastric catheter
* Heart and lung transplant
* Increase in PIC
* Refusal of the parents or legal guardian
* Enrolment in other research protocols

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Asynchrony Index | 60 minutes of each ventilatory trial, PSV or NAVA

SECONDARY OUTCOMES:
Arterial blood gases | End of each ventilatory trial

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Chidini, MD, Principal Investigator — Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico; Calderini Edoardo, MD, Study Chair — Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico; Giorgio Conti, MD, Phd, Study Chair — University Sacred Heart, Rome
Locations (1):
- Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] 1) Colombo D, Cammarota G, Bergamaschi V, De Lucia M, Corte FD, Navalesi P. Physiologic response to varying levels of pressure support and neurally adjusted ventilatory assist in patients with acute respiratory failure. Intensive Care Med 2008;34:2010-2018. 2) Sinderby C, Navalesi P, Beck J, Skrobik Y, Comtois N, Friberg S, Gottfried SB, Lindstrom L. Neural control of mechanical ventilation in respiratory failure. Nat Med 1999;5:1433-1436. 3) Sinderby C, Beck J, Spahija J, de Marchie M, Lacroix J, Navalesi P, Slutsky AS. Inspiratory Muscle Unloading by Neurally Adjusted Ventilatory Assist during Maximal Inspiratory Efforts in Healthy Subjects. Chest 2007;131:711-717. 4) Beck J, Brander L, Slutsky AS, Reilly MC, Dunn MS, Sinderby C. Non-invasive neurally adjusted ventilatory assist in rabbits with acute lung injury. Intensive Care Med 2008;34:316-323